CLINICAL TRIAL: NCT00519870
Title: Losartan Decreases Pulmonary Artery Pressure and Improves Exercise Capacity in Patients With Pulmonary Hypertension
Brief Title: Losartan Therapy in Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA04/127
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Angiotensin receptor blocker; Calcium channel blocker
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Nifedipine; Losartan

ARMS (1):
- I, II (Active Comparator): I: nifedipine II: losartan
  Interventions: Drug: nifedipine, losartan; Drug: losartan

INTERVENTIONS:
Drug: nifedipine, losartan — I: nifedipine 30 mg/d II: losartan 50 mg/d
  Other Names: nifedipine (Adalat Crono, Bayer AG, Leverkusen, Germany); losartan (Cozaar, Merck Sharp & Dohme, Wilmington, DE, USA)
Drug: losartan — II: losartan
  Other Names: losartan (Cozaar, Merck Sharp & Dohme, Wilmington, DE, USA) 50 mg/d
Drug: Nifedipine, losartan — I: nifedipine II: losartan

SUMMARY:
In addition to being effective vasodilators, angiotensin-converting enzyme inhibitors (ACEIs) and angiotensin receptor blockers (ARBs) exert neurohumoral inhibitory actions, such as the inhibition of vascular remodeling and smooth muscle cell proliferation and the amelioration of endothelial dysfunction. These beneficial effects, render those agents appropriate for use in the treatment of pulmonary hypertension. However, data regarding the use of ACEIs or ARBs in the treatment of PHT are limited. In this study, efficacy of an ARB, losartan was compared with those of the calcium channel blocker, nifedipine in the treatment of pulmonary hypertension using echocardiographic, 6-minute walk test (6MWT), cardiopulmonary exercise test, and endothelin-1 levels.Losartan is as effective as nifedipine for reducing Doppler echocardiographically measured PAP and improving exercise capacity on 6MWT and CPET. However the short-term use of losartan or nifedipine had no statistically significant effect on endothelin-1 levels in patients with PHT.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension diagnosed by Doppler echocardiographic examination (a mean pulmonary artery pressure of > 26mmHg)

Exclusion Criteria:

* acute infectious or inflammatory disease,
* exacerbation of chronic obstructive pulmonary disease,
* malignancy,
* acute coronary syndrome in the last 4 weeks,
* uncontrolled arrhythmia and hypertension,
* decompensated heart failure,
* acute pulmonary emboli,
* thrombus in a lower extremity,
* oxygen saturation below 85% at rest,
* failure to cooperate with CPET

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Serife Savas Bozbas, MD, Principal Investigator — Baskent University Faculty of Medicine, Department of Pulmonary Disease; Fusun Oner Eyuboglu, MD, Study Chair — Baskent University Faculty of Medicine, Department of Pulmonary Disease